CLINICAL TRIAL: NCT04029324
Title: Clinical Outcomes of Immediate Implant Placement and Early Implant Placement: a Randomized Controlled Clinical Trial
Brief Title: Clinical Outcomes of Immediate Implant Placement and Early Implant Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Junyu Shi, Principal investigator, clinical professor,Department of Implant Dentistry, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 136-2019
Record Dates: First submitted 2019-07-07; First posted 2019-07-23 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Tooth Fractures; Tooth Diseases
MeSH Terms: conditions — Tooth Fractures; Tooth Diseases | interventions — Tooth Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate implant placement (Active Comparator): Implants are placed immediately after extraction
  Interventions: Procedure: tooth extraction; Procedure: Implant placement; Procedure: Bone augmentation
- Early implant placement (Placebo Comparator): Implants are placed 4-8 weeks after extraction
  Interventions: Procedure: tooth extraction; Procedure: Implant placement; Procedure: Bone augmentation; Procedure: Coronally repositioned flap

INTERVENTIONS:
Procedure: tooth extraction — Under local anesthesia, tooth will be extracted atraumatically.
Procedure: Implant placement — Dental implants will be placed according to the instructions in fresh sockets or alveolar ridge.
Procedure: Bone augmentation — Bone substitute will be used to augment or maintain the bone contour.
Procedure: Coronally repositioned flap — After periosteal releasing incision, mucoperiosteal flap will be sutured at a more coronally position
  Arms: Early implant placement

SUMMARY:
Immediate implant placement (IIP) has been an attractive treatment concept for both patients and clinicians due to reduced surgical interventions and total treatment span. Although soft-tissue alterations or midfacial recession have been demonstrated in previous studies, recent studies have reported positive result following IIP with the modification of surgical interventions. However, high-quality evidence (≥Ib: evidence from at least one randomized controlled trial) on comparing the clinical outcome of IIP with early implant placement (type 2) is limited.

ELIGIBILITY:
Inclusion Criteria:

* age ≧18 years
* single hopeless teeth in anterior maxilla
* enough apical bone volume to achieve primary stability (>4mm)

Exclusion Criteria:

* active periodontoal infection
* incomplete buccal bone plate
* unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Midfacial recession | 1-year follow-up
  Recession of midfacial gingival level before extraction and 1-year follow-up

SECONDARY OUTCOMES:
Papillae recession | 1-year follow-up
  Recession of papillae before extraction and 1-year follow-up
marginal bone loss | 1-year follow-up
  marginal bone level between crown delivery and 1-year follow-up
Probing depth | T2:crown delivery, T3: 1-year follow-up
  Probing depth between crown delivery and 1-year follow-up
Bleeding on probing % | T2:crown delivery, T3: 1-year follow-up
  Bleeding on probing % between crown delivery and 1-year follow-up
Pink esthetic score | T2:crown delivery, T3: 1-year follow-up
Visual Analogue Scale assessement | T1: immediately after surgery,T2:crown delivery, T3: 1-year follow-up
  Visual Analogue Scale on post-operative pain, esthetics and function

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai NinthPeoples' Hospital, Shanghai, China